CLINICAL TRIAL: NCT05105867
Title: A Single-Arm, Open-Label Study to Evaluate the Efficacy and Safety of Anti-CD19 Universal CAR-T Cells in the Treatment of CD19+ Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia and Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: CD19 Targeted Universal Chimeric Antigen Receptor T Cells Injection for CD19+ Refractory/Relapsed B-cell Malignancies
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Collaborators: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry); Kunming Hope of Health Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC011-411
Record Dates: First submitted 2021-10-25; First posted 2021-11-03 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-04

CONDITIONS: Relapsed or Refractory B-cell Acute Lymphoblastic Leukemia; Relapsed or Refractory B-cell Non-hodgkin Lymphoma
MeSH Terms: conditions — Recurrence; Burkitt Lymphoma; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-CD19 Universal CAR-T Cells injection (Experimental): Anti-CD19 Universal CAR-T Cells injection will be administered by vein after lymphodepletion .
  Interventions: Biological: Anti-CD19 Universal CAR-T Cells injection

INTERVENTIONS:
Biological: Anti-CD19 Universal CAR-T Cells injection — Anti-CD19 Universal CAR-T Cells injection will be administered by vein after lymphodepletion.

SUMMARY:
It is a single-arm, open-label clinical study to assess the safety and efficacy of the Anti-CD19 Universal CAR-T Cells injection for patients with CD19+ refractory/relapsed B cell acute lymphoblastic leukemia and B cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
The study consists of the following periods: screening, lymphodepletion, CAR-T cell infusion, safety follow up, and long term follow-up.

ELIGIBILITY:
Key Inclusion Criteria:

1. Eastern Cooperative Oncology Group Performance Status of 0 or 1；
2. Expected survival time ≥12 weeks;
3. Adequate hematological, renal and liver function;
4. Subjects understand and voluntarily sign the informed consent form.

Key Exclusion Criteria:

1. Positive for any of the following etiological tests: HIV, HBV, HCV, TPPA ;
2. Cyclophosphamide or fludarabine is contraindicated for subjects ;
3. Active central nervous system (CNS) involvement by malignancy；
4. Active infection.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicities | Up to 4 weeks after CAR-T infusion
  Incidence of dose-limiting toxicities as protocol-defined

SECONDARY OUTCOMES:
Objective response rate (ORR) | At 4,12,24 weeks after CAR-T infusion
  Objective response rate after CAR-T infusion

CONTACTS AND LOCATIONS:
Overall Officials: Sanbin Wang, Professor, Principal Investigator — 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China
Locations (1):
- 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China, Kunming, Yunnan, China